CLINICAL TRIAL: NCT02459236
Title: A Randomized, Double-Blind, Placebo-Controlled Study of Intermittent Doses of CERC-301 in the Treatment of Subjects With Severe Depression Despite Antidepressant Treatment
Brief Title: A Study of Intermittent Doses of CERC-301 in MDD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Avalo Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Clin301-203
Record Dates: First submitted 2015-05-27; First posted 2015-06-02 (Estimated); Last update posted 2017-09-28 (Actual); Status verified 2017-09

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- CERC-301 12mg (Experimental): The study includes two dose administrations 7 days apart (Day 0 and Day 7) followed by 14 days of observation for a total of 21 days.
  Interventions: Drug: CERC-301
- CERC-301 20mg (Experimental): The study includes two dose administrations 7 days apart (Day 0 and Day 7) followed by 14 days of observation for a total of 21 days.
  Interventions: Drug: CERC-301
- Placebo (Placebo Comparator): The study includes two dose administrations 7 days apart (Day 0 and Day 7) followed by 14 days of observation for a total of 21 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CERC-301 — CERC-301, a highly selective, orally bioavailable, NMDA receptor subunit 2B (NR2B), also referred to as Glutamate NMDA receptor subunit epsilon-2 (GluN2B) antagonist
  Arms: CERC-301 12mg; CERC-301 20mg
Drug: Placebo
  Arms: Placebo

SUMMARY:
There is a significant unmet medical need for rapidly acting treatment of subjects with severe major depressive disorder (MDD) who have not adequately responded to antidepressant therapy. Alternative therapies require weeks to achieve full efficacy, may have significant side effects, and still fail in a high percentage of subjects. Rapid reduction of severe depression by pharmacological therapy is important to reduce the need for hospitalization and risk of self-harm and mortality. CERC-301, a highly selective, orally bioavailable, N-methyl-D-aspartate (NMDA) receptor subunit 2B (NR2B), also referred to as Glutamate NMDA receptor subunit epsilon-2 (GluN2B) antagonist, would be a therapeutic breakthrough if it provides rapid onset of antidepressant effects and an effect size similar to that seen with experimental intravenous NMDA modulators.

DETAILED DESCRIPTION:
The study will evaluate the antidepressant effect of one or two administrations of two doses of CERC-301 (12 mg and 20 mg) in subjects with MDD who are currently experiencing a severe depressive episode despite stable ongoing treatment with a selective serotonin- or serotonin-norepinephrine reuptake inhibitor (SSRI or SNRI).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of MDD recurrent without psychotic features according to DSM-IV-TR criteria with diagnosis confirmed using the Structured Clinical Interview for DSM-IV Axis I Disorders Clinical Trials Version (SCID-CT).
2. Lifetime history of ≥2 major depressive episodes, for which at least one required treatment with SSRI or SNRI antidepressants.
3. History during the current major depressive episode of failure to achieve a satisfactory response (e.g., less than 50% improvement of depression symptoms) to ≤3 treatment courses of a therapeutic dose of an antidepressant therapy of at least 8 weeks duration during the current episode, according to the Massachusetts General Hospital Antidepressant Treatment Response Questionnaire.

Exclusion Criteria:

1. Duration of current depression episode ≥2 years or diagnosis of Persistent Depressive Disorder (DSM-V) or Dysthymic Disorder (DSM-IV)
2. Use of other NMDA-receptor modulators (e.g., dextromethorphan, ketamine, amantadine, memantine) within 30 days of screening and throughout the study.
3. History of use of an NMDA-receptor modulator for the treatment of MDD.
4. Use of bupropion, tricyclic antidepressants, antipsychotics, stimulants, or lithium within 8 weeks prior to screening
5. Initiation of psychotherapy or a change in intensity of psychotherapy or other non-drug therapies (e.g., hypnosis, acupuncture) within 8 weeks prior to screening.
6. Electroconvulsive therapy, transcranial magnetic stimulation, or vagal nerve stimulation during the current depressive episode.
7. Excessive alcohol use, which is defined by the Centers for Disease Control as >1 drink per day for women and >2 drinks per day for men.
8. Current diagnosis of a Substance Use (including alcohol) Disorder (Abuse or Dependence, as defined by DSM-IV/V), with the exception of nicotine dependence, at screening or within 6 months prior to screening.
9. Active, comorbid disease that might limit the ability of the subject to participate in the study as determined by the Investigator (i.e., poorly controlled diabetes mellitus, congestive heart failure, etc.).
10. Current neurologic or neuropsychiatric disorder which could interfere with the ability to diagnose or assess MDD or which could cause or contribute to depressive symptomatology (e.g., Alzheimer's disease, Parkinson's diseases, chronic pain syndromes, including fibromyalgia, substance use disorder, post-partum depression).
11. Lifetime history of the following disorders: Bipolar I, II, or Not Otherwise Specified (NOS) mood disorders, eating disorders , schizophrenia and other psychotic disorders, sleep disorders , significant cognitive disorders, dissociative disorders, impulse control disorders, and borderline, antisocial, paranoid, schizoid, schizotypal, or histrionic personality disorders.
12. Subjects with suicidal behavior within 6 months prior to screening as measured by the Columbia-Suicide Severity Rating Scale (C-SSRS) "Baseline/Screening" version.
13. Elevated seated blood pressure at screening and prior to randomization
14. Lifetime history of stroke or congestive heart failure, atrial fibrillation or coronary artery disease.
15. Clinically significant current liver disease or liver enzyme (GGT, ALT, AST, total bilirubin) elevations at screening above 2 × the ULN.
16. Clinically significant renal impairment defined as estimated creatinine clearance [CrCl] <50 mL/min at screening measured using Cockcroft-Gault formula.
17. Fasting serum glucose >140 mg/dL.
18. Subjects who, in the opinion of the Investigator, are not appropriate for a 21-day placebo-controlled study due to risk of significant threat to self or others during screening or study conduct.
19. Previous participation in an investigational study using CERC-301.
20. Participation in an investigational drug or device study within the 6 months prior to screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2015-06; Primary Completion 2016-09 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in Bech-6 from baseline | average of 2 and 4 days post-treatment
  To evaluate the antidepressant effect of CERC-301 (12 or 20 mg) compared to placebo averaged between 2 and 4 days post-treatment with study drug assessed by the 6-item unidimensional subset (Bech-6) of the 17-item Hamilton Depression Rating Scale (HDRS-17)

SECONDARY OUTCOMES:
Change from baseline in Santen-7 | averaged between 2 and 4 days post treatment
  To evaluate the antidepressant effect of a single dose of CERC-301 (12 or 20 mg) compared to placebo averaged between 2 and 4 days post-treatment with study drug assessed by the 7-item unidimensional subset of the HDRS-17, the Santen-7
Change from baseline in HDRS-17 | averaged between 2 and 4 days post treatment
  To evaluate the antidepressant effect of a single dose of CERC-301 (12 or 20 mg) compared to placebo averaged between 2 and 4 days post-treatment with study drug assessed by the HDRS-17
Change from baseline in Bech-6 | 2, 4, 7 days after each dose, and 14 days after last dose of study drug treatment
  To evaluate the antidepressant effect of CERC-301 at 2, 4, 7 days after each dose, and 14 days after last dose of study drug treatment assessed by the Bech-6.
Change from baseline in Santen-7 | 2, 4, 7 days after each dose, and 14 days after last dose of study drug treatment
  To evaluate the antidepressant effect of CERC-301 at 2, 4, 7 days after each dose, and 14 days after last dose of study drug treatment assessed by the Santen-7.
Change from baseline in HDRS-17 | 2, 4, 7 days after each dose, and 14 days after last dose of study drug treatment
  To evaluate the antidepressant effect of CERC-301 at 2, 4, 7 days after each dose, and 14 days after last dose of study drug treatment assessed by the HDRS-17.
Change from baseline in CUDOS-A | 2, 4, 7 days after each dose, and 14 days after last dose of study drug treatment
  To evaluate the antidepressant effect of CERC-301 at 2, 4, 7 days after each dose, and 14 days after last dose of study drug treatment assessed by the Clinically Useful Depression Outcome Scale-Anxiety (CUDOS-A).
Change from baseline in SHAPS-SR | 2, 4, 7 days after each dose, and 14 days after last dose of study drug treatment
  To evaluate the antidepressant effect of CERC-301 at 2, 4, 7 days after each dose, and 14 days after last dose of study drug treatment assessed by the Snaith-Hamilton Pleasure Scale Self Report (SHAPS-SR)
Change from baseline in QIDS-SR | 7 days after each dose and 14 days after last dose of study drug treatment
  To evaluate the antidepressant effect of CERC-301 at 7 days after each dose and 14 days after last dose of study drug treatment assessed by the Quick Inventory of Depressive Symptomatology Self Report (QIDS-SR)
Change from baseline in CGI-I | 7 days after each dose and 14 days after last dose of study drug treatment
  To evaluate the antidepressant effect of CERC-301 at 7 days after each dose and 14 days after last dose of study drug treatment assessed by the Clinical Global Impression-Improvement (CGI-I)
Change from baseline in CGI-S | 7 days after each dose and 14 days after last dose of study drug treatment
  To evaluate the antidepressant effect of CERC-301 at 7 days after each dose and 14 days after last dose of study drug treatment assessed by the Clinical Global Impression -Severity (CGI-S)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald N Marcus, MD, Study Director — Avalo Therapeutics, Inc.
Locations (13):
- United States (13):
  - Pharmacology Research Institute (PRI), Newport Beach, California
  - Institute for Advanced Medical Research, Alpharetta, Georgia
  - Chicago Research Center, Inc., Chicago, Illinois
  - Alexian Brothers Center for Psychiatric Research, Hoffman Estates, Illinois
  - Psychiatric Care and Research Center, O'Fallon, Missouri
  - Bioscience Research LLC, Mount Kisco, New York
  - The Medical Research Network, LLC, New York, New York
  - Fingerlakes Clinical Research, Rochester, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - Summit Research Network (Oregon) Inc., Portland, Oregon
  - Lehigh Center for Clinical Research, Allentown, Pennsylvania
  - Research Strategies of Memphis, LLC, Memphis, Tennessee
  - Northwest Clinical Research Center, Bellevue, Washington